CLINICAL TRIAL: NCT07040722
Title: Effects of the Use of an Immersive Virtual Reality Device on Handwriting in Children Aged 6 to 13 With Handwriting Difficulties : a Randomized Multiple Baseline Single-case Experimental Design (SCED)
Brief Title: Effects of the Use of an Immersive Virtual Reality Device on Handwriting in Children Aged 6 to 13 With Handwriting Difficulties ( RVALIGO )
Acronym: RVALIGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ildys (Other)
Collaborators: LP3C, University of Brest (Unknown); LaTim Laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RI2024_020
Record Dates: First submitted 2025-05-06; First posted 2025-06-27 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-06

CONDITIONS: Children With a Need of Rehabilitation for Handwriting
Keywords: Handwriting difficulties; Virtual reality; SCED; Children; Pediatric rehabilitation
MeSH Terms: interventions — BaseLine dental cement; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with handwriting difficulties (Experimental): Children included in the study will carry out the baseline (i.e. a 'control' phase) as well as the intervention (corresponding to the introduction of the VR)
  Interventions: Other: Baseline; Other: Intervention

INTERVENTIONS:
Other: Baseline — During the baseline, children will carry out their standard paper-and-pencil exercises for writing difficulties (that their perform during usual rehabilitation).
Other: Intervention — During the intervention, they will carry out usual exercises and they will use VR 15 minutes during each session

SUMMARY:
Difficulties in learning to write affect a large number of children and can have a significant impact on their personal and professional future. To facilitate this learning process, develop fun, motivating and effective devices for the different skills involved in writing (motor skills, postural control, visual attention, letter recognition) is needing. Virtual Reality (VR) seems to be a promising tool for this purpose.

The SCED (Single Case Experimental Design) methodology is adapted to this study to evaluate the impact of VR on learning to write, as it allows a high level of evidence and is applicable to a heterogeneous population such as that affected by difficulties in learning to write. The study will include an original study of 3 children and 3 replications of 3 children each. In total, 12 children will be included in four different settings. This study will determine whether VR training can facilitate learning to write.

The main objective of this study is to evaluate the impact of immersive virtual reality training on handwriting using the Evaligo tool to assess static, kinematic and pressure parameters of handwriting in children aged 6 to 13 with handwriting difficulties according to a SCED methodology.

DETAILED DESCRIPTION:
5% to 30% of children in mainstream education experience difficulties with writing acquisition. This prevalence increases among children with motor disabilities such as cerebral palsy, coordination disorders, or attention-deficit/hyperactivity disorder. Writing difficulties can significantly impact other core learning areas, as well as children's development and future (e.g., increased risk of academic failure, reduced access to higher education, lower self-esteem).

These writing difficulties are multifactorial and require individualized intervention. Fine motor skills, postural control, and visual attention-key abilities in the learning of writing-are often impaired in children with writing difficulties.

Virtual reality (VR) can be defined as the digital simulation of a virtual environment with which users can interact through their own movements. In immersive VR, users wear a head mounted display (HMD) that allows them to be fully immersed in the virtual environment.

VR has been shown to improve upper limb function and postural control in pediatric rehabilitation. It integrates several features that support motor learning, including task repetition, sensory feedback, and enhanced motivation during exercises.

Using VR training to target skills associated with writing thus appears to be relevant. Furthermore, proposing writing training through gross motor activities in VR may facilitate the consolidation of motor programs necessary for letter formation.

This engaging system could increase the amount of training, introduce variability between virtual and real-world practice, and promote the child's autonomy-all key elements for effective learning and, consequently, improved writing skills.

The following hypotheses are proposing:

* Immersive VR training will facilitate the learning of writing.
* Skills associated with writing (visual attention, fine motor skills, gross motor skills, postural control, and letter recognition) will be improved through immersive VR training.
* Motivation will be maintained throughout the intervention due to the use of VR.

A multicentre, multiple baseline SCED, following the SCRIBE recommendations will be conducting. This is a prospective design allowing intensive study of one or a few individuals with the aim of measuring their state (baseline) and the state engendered by a therapeutic intervention. It is the demonstration of 3 effects that allows us to conclude that the intervention is effective (for example: measurement of 3 effects in 3 different patients, effects corresponding to the introduction of the therapeutic intervention). This design is suitable because i/ each subject is his or her own control, which makes it possible to avoid matching difficulties (complex in our case, given the varied expected profiles of children with writing disorders) and to respect the individualised nature of the treatment, ii/ it allows the inclusion of a small number of subjects, which is well suited to a pilot study, iii/ the repeated measurements of the main outcome make it possible to ensure that the changes observed are indeed linked to the intervention. This design is adapted to the specificities of rehabilitation treatment, with an effect that lasts over time.

In this study, baseline will be randomised for each child. It will last from 2 to 6 weeks (6 to 14 sessions of repeated measurements of the primary endpoint), starting at visit 1. From this phase onwards, the children will benefit from an intervention ('control', i.e. the usual care of the child by the usual therapist) aimed at training writing (paper/pencil).

The therapeutic intervention (introduction of the VR HMD) will last 8 weeks (16 sessions of repeated measures of the primary endpoint). It will include 2 intervention sessions with the child's usual care therapist per week (during which the repeated measures of the primary endpoint will be performed by the child's therapist).

Inclusion visits (V1), visits at the start of the intervention (V2), and visits at the end of the intervention (V5) will be used to assess the skills associated with writing. V3 and V4 will evaluate the sense of presence of children just after the use of the HMD.

ELIGIBILITY:
Inclusion Criteria:

* Age : 6-13 years
* BHK: degradation score ≥ 1 standard deviation. The BHK will be administered at the time of the inclusion visit (V1) and/or child with writing difficulties in in daily activities.
* Children benefiting or to benefit from rehabilitation care to improve handwriting skills.
* Be able to understand instructions and complete all assessments.

Exclusion Criteria:

* Contraindications to using a virtual reality HMD
* Severe visual impairment
* Facial injury
* Epilepsy
* Lack of parental and/or child consent

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of immersive virtual reality training on learning using the Evaligo score. | This score will be assessed twice a week during the baseline and intervention periods (10 to 14 weeks depending on the baseline).
  The Evaligo score assesses static, kinematic and pressure parameters of handwriting in children aged 6 to 13 with handwriting learning difficulties, using a SCED methodology.
  This assessment has several advantages in this study design: its validity has been verified, it can be repeated a large number of times without test-retest effect, it is sensitive to change and is quick to set up (around 5 minutes), which reduces the burden of assessments for the participating children and therapists.
  • This score is obtained on the basis of a brief evaluation of around 5 minutes (and repeated, according to the SCED methodology) of trained items (during the intervention), throughout participation in the research (baseline, intervention).
  The minimum score is 0 (worst), the maximum score is 1 (best).

SECONDARY OUTCOMES:
Assess fine and gross motor skills | This criterion will be measured (during the first week of the baseline), during the first week of intervention (V2), and the visit at the 8th of the inetervention (V5)
  Evolution of the score of the Bruininks-Oseretsky Test of Motor Proficiency Brief Form. This test has been validated in a population aged 4 to 21 years. It assesses gross and fine motor skills. The strength subtest will be our control measure in this SCED. The control measure will make it possible to assess an untrained parameter (in this case strength), which is supposed to remain stable during the intervention.
  The maximum score for fine motor skills part is 60, the minimum score is 0. A high score means high performance in fine motor skills.
  The maximum score for gross motor skills part is 65, the minimum score is 0. A high score means high performance in gross motor skills.
Assess visual attention | The criterion will be measured during the first week of the baseline, during the first week of intervention (V2), and the visit at the 8th of the intervention (V5).
  Evolution of the score of the sky search and geographic map subtests of the Test of Everyday Attention for Children (TEA-CH). It assesses visual attention. This test has been validated in a population aged 6 to 16 years. Two subtest will be used: "Map Mission" and "Sky Search" in this study.
  The maximum score for Map Mission subtest is 80, the minimum score is 1. A high score means high performance in visual attention. The maximum raw score for Sky Search is 20, the minimum score is 1. A high score means high performance in visual attention.
Assess postural control | The criterion will be measured during the first week of the baseline, during the first week of intervention (V2), and the visit at the 8th of the intervention (V5).
  Evolution of the Pediatric Reach Test (PRT) score, validated in children aged 5 to 15 with or without motor disorders. This test assesses postural control. The score is the difference, in cm, between the starting position and the finishing position.
Determine whether a generalization of learning to write takes place on the paper/pencil writing activity. | The BHK will be taken at the first week of the baseline and at the 8th week of the intervention (V5).
  Evolution of the BHK score, the benchmark test for assessing handwriting. In the BHK (Brave Handwriting Kindergarten), the child is asked to copy a text for 5 minutes. Blind double scoring is used (the scorer does not know when the child has copied the text). A degradation score is calculated: the higher the score, the more "degraded" the quality of the child's handwriting. The standardized score is taken into account for inclusion (to situate the child's performance in relation to his class), while the raw score is taken into account over the course of the intervention (allowing comparison of the subject with himself).
  The maximum score for the handwriting quality is 65. A high score means low performance in handwriting.
Check that the child's motivation is maintained during training. | Analog scale score at the end of each session, during baseline and intervention (10 to 14 weeks depending on the baseline).
  Visual analogue scale score at each end of session, during baseline and intervention. The maximum score is 10, the minimum score is 0. A high score means a high motivation during session.
Assess satisfaction with the intervention : CSQ-8 | Assessment carried out at the 8th week of the intervention.
  The CSQ-8 is a questionnaire used to assess customer satisfaction. The families of the children who took part in the study will be invited to complete this questionnaire during the V5 visit. This questionnaire has been adapted for different populations (families).
  Scores range from 8 to 32, higher values indicates higher satisfaction.
Assess satisfaction with the intervention | Evaluation carried out at 8th week of the intervention.
  A visual analogue scale (VAS) will be implemented during the V5 visit to determine children's and professionals' satisfaction with the use of the immersive VR headset. The maximum score is 10, the minimum score is 0. A high score means a high global satisfaction during the study.
Evaluate the usability of the solution | Evaluation carried out at 8th week of the intervention
  SUS (System Usability Scale) questionnaire to be completed by children and professionals.
  This questionnaire is currently the most widely used in the scientific community for measuring user satisfaction with a product, interactive system or service.
  Scores range from 0 to 100, higher values indicates higher satisfaction.
Assess the child's sense of presence in the virtual environment | Evaluation carried out at the first session of the intervention phase (Session 1 of the intervention phase), and at the last session pf the intervention phase (Session 16 of the intervention phase).
  Spatial Presence for Immersive Environments questionnaire (SP-IE), to be completed by the children to assess their sense of presence in the virtual environment. The SP-IE comprises 20 items.
  Each item is assessed on a 5-point Likert Scale, ranging from 1 (strongly disagree) to 5 (strongly agree)
Assessing language levels : letter recognition | The language levels will be measured during the first week of the baseline, during the first week of intervention (V2), and the visit at the 8th of the intervention (V5)
  Evolve assessments of language skills into assessments that are used as references in teaching with letter recognition. For the subtest letter recognition, the maximum score is 6 and the minimum score is 0.
Assessing language levels : knowledge of letter names | The language levels will be measured during the first week of the baseline, during the first week of intervention (V2), and the visit at the 8th of the intervention (V5)
  Evolve assessments of language skills into assessments that are used as references in teaching with knowledge of letter names. For the subtest knowledge of letters names, the maximum score is 12, and the minimum score is 0.
Assessing language levels : writing a letter | The language levels will be measured during the first week of the baseline, during the first week of intervention (V2), and the visit at the 8th of the intervention (V5)
  Evolve assessments of language skills into assessments that are used as references in teaching with writing a letter. For the subtest writing a letter, the maximum score is 12 and the minimum score is 0.
Assessing language levels : recognition of allographs | The language levels will be measured during the first week of the baseline, during the first week of intervention (V2), and the visit at the 8th of the intervention (V5)
  Evolve assessments of language skills into assessments that are used as references in teaching with recognition of allographs. For the subtest recognition of allographs, the maximum score is 6 and the minimum score is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Jéromine HERVO, Coordinator Investigator, Principal Investigator — Fondation Ildys
Locations (5):
- France (5):
  - Cabinet d'ergothérapie Scol'Ergo, Pont-de-l'Arche, Eure
  - Cabinet Ker ergo, Brest, Finistère
  - Fondation ILDYS, Brest, Finistère
  - Cabinet d'ergothérapie - Maison des Korrigans, Lesneven, Finistère
  - Fondation ILDYS, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapp C, Perlini T, Baggio S, Stephan P, Urrego AR, Rengade CE, Macias M, Hainard N, Halfon O. [Psychometric properties of the Consumer Satisfaction Questionnaire (CSQ-8) and the Helping Alliance Questionnaire (HAQ)]. Sante Publique. 2014 May-Jun;26(3):337-44. French. PMID 25291882
- [Background] Bartlett D, Birmingham T. Validity and reliability of a pediatric reach test. Pediatr Phys Ther. 2003 Summer;15(2):84-92. doi: 10.1097/01.PEP.0000067885.63909.5C. PMID 17057438
- [Background] Manly T, Anderson V, Nimmo-Smith I, Turner A, Watson P, Robertson IH. The differential assessment of children's attention: the Test of Everyday Attention for Children (TEA-Ch), normative sample and ADHD performance. J Child Psychol Psychiatry. 2001 Nov;42(8):1065-81. doi: 10.1111/1469-7610.00806. PMID 11806689
- [Background] Krasny-Pacini A, Evans J. Single-case experimental designs to assess intervention effectiveness in rehabilitation: A practical guide. Ann Phys Rehabil Med. 2018 May;61(3):164-179. doi: 10.1016/j.rehab.2017.12.002. Epub 2017 Dec 15. PMID 29253607
- [Background] Tate RL, Perdices M, Rosenkoetter U, Shadish W, Vohra S, Barlow DH, Horner R, Kazdin A, Kratochwill T, McDonald S, Sampson M, Shamseer L, Togher L, Albin R, Backman C, Douglas J, Evans JJ, Gast D, Manolov R, Mitchell G, Nickels L, Nikles J, Ownsworth T, Rose M, Schmid CH, Wilson B. The Single-Case Reporting Guideline In BEhavioural Interventions (SCRIBE) 2016 Statement. Phys Ther. 2016 Jul;96(7):e1-e10. doi: 10.2522/ptj.2016.96.7.e1. PMID 27371692
- [Background] Bara F, Bonneton-Botte N. Learning Letters With the Whole Body: Visuomotor Versus Visual Teaching in Kindergarten. Percept Mot Skills. 2018 Feb;125(1):190-207. doi: 10.1177/0031512517742284. Epub 2017 Nov 21. PMID 29161949
- [Background] Tatla SK, Sauve K, Virji-Babul N, Holsti L, Butler C, Van Der Loos HF. Evidence for outcomes of motivational rehabilitation interventions for children and adolescents with cerebral palsy: an American Academy for Cerebral Palsy and Developmental Medicine systematic review. Dev Med Child Neurol. 2013 Jul;55(7):593-601. doi: 10.1111/dmcn.12147. Epub 2013 Mar 29. PMID 23550896
- [Background] Warnier N, Lambregts S, Port IV. Effect of Virtual Reality Therapy on Balance and Walking in Children with Cerebral Palsy: A Systematic Review. Dev Neurorehabil. 2020 Nov;23(8):502-518. doi: 10.1080/17518423.2019.1683907. Epub 2019 Nov 1. PMID 31674852
- [Background] Burin-Chu S, Baillet H, Leconte P, Lejeune L, Thouvarecq R, Benguigui N. Effectiveness of virtual reality interventions of the upper limb in children and young adults with cerebral palsy: A systematic review with meta-analysis. Clin Rehabil. 2024 Jan;38(1):15-33. doi: 10.1177/02692155231187858. Epub 2023 Jul 27. PMID 37499213
- [Background] Monge Pereira E, Molina Rueda F, Alguacil Diego IM, Cano de la Cuerda R, de Mauro A, Miangolarra Page JC; CONSOLIDER-Ingenio 2010. Use of virtual reality systems as proprioception method in cerebral palsy: clinical practice guideline. Neurologia. 2014 Nov-Dec;29(9):550-9. doi: 10.1016/j.nrl.2011.12.004. Epub 2012 Feb 17. English, Spanish. PMID 22341675
- [Background] Adamovich SV, Fluet GG, Tunik E, Merians AS. Sensorimotor training in virtual reality: a review. NeuroRehabilitation. 2009;25(1):29-44. doi: 10.3233/NRE-2009-0497. PMID 19713617
- [Background] Lopez C, Vaivre-Douret L. Influence of visual control on the quality of graphic gesture in children with handwriting disorders. Sci Rep. 2021 Dec 7;11(1):23537. doi: 10.1038/s41598-021-02969-7. PMID 34876643
- [Background] Bumin G, Kavak ST. An investigation of the factors affecting handwriting skill in children with hemiplegic cerebral palsy. Disabil Rehabil. 2010;32(8):692-703. doi: 10.3109/09638281003654789. PMID 20205584
- [Background] Biotteau M, Danna J, Baudou E, Puyjarinet F, Velay JL, Albaret JM, Chaix Y. Developmental coordination disorder and dysgraphia: signs and symptoms, diagnosis, and rehabilitation. Neuropsychiatr Dis Treat. 2019 Jul 8;15:1873-1885. doi: 10.2147/NDT.S120514. eCollection 2019. PMID 31371960
- [Background] Overvelde A, Hulstijn W. Handwriting development in grade 2 and grade 3 primary school children with normal, at risk, or dysgraphic characteristics. Res Dev Disabil. 2011 Mar-Apr;32(2):540-8. doi: 10.1016/j.ridd.2010.12.027. Epub 2011 Jan 26. PMID 21269805
- [Background] Bonneton-Botte N, Miramand L, Bailly R, Pons C. Teaching and Rehabilitation of Handwriting for Children in the Digital Age: Issues and Challenges. Children (Basel). 2023 Jun 22;10(7):1096. doi: 10.3390/children10071096. PMID 37508593